CLINICAL TRIAL: NCT06331689
Title: EPIDEMIOLOGY AND ITS RESULTS IN HIP FRACTURES FOLLOWED IN POSTOPERATIVE INTENSIVE CARE
Acronym: Hip fractures
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Yıldız, Assistant Professor, Kutahya Health Sciences University
Other Study IDs: hipksbu1234
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Hip Fracture; Mortality Rate
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mortality ratio — Mortality rates at 30-day, 90-day and 1-year intervals

SUMMARY:
Type of study: Observational study Goal of this : We conducted a retrospective evaluation of patients with HF who received postoperative ICU, with a focus on 30-day, 90-day and 1-year mortality outcomes.

Participant population/health conditions:Patients over the age of 18 who are hospitalized in the intensive care unit of our hospital after hip fracture operation.

DETAILED DESCRIPTION:
The proportion of elderly individual aged 65 and over in the global populatin is currently %9 and hip fractures (HFs) are a leading injury in this population worldwide. We conducted a retrospective evaluation of patients with HF who received postoperative ICU, with a focus on 30-day, 90-day and 1-year mortality outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with postoperative hip fractures hospitalized in the intensive care unit of our hospital

Exclusion Criteria:

* Patients who do not have a hip fracture operation will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with postoperative hip fractures in intensive care
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
mortalite ratio | one year
  Patients with hip fracture who received postoperative intensive care unit , with a focus on 30-day, 90-day and 1-year mortality outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL YILDIZ, Ass. Prof., Study Director — Kutahya HSU
Locations (2):
- Turkey (Türkiye) (2):
  - Kutahya Health Sciences University, Kütahya
  - Kütahya Health Sciences University, Kütahya

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19335921/